CLINICAL TRIAL: NCT03594474
Title: Does Early Higher Intravenous Lipid Intake Decrease Weight Loss in Very Low Birth Weight Infants?
Brief Title: Early Higher Intravenous Lipid Intake in VLBW Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Belal Alshaikh (Other)
Responsible Party: Sponsor-Investigator, Belal Alshaikh, Neonatologist, University of Calgary
Organization: University of Calgary (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB17-2236
Record Dates: First submitted 2018-07-09; First posted 2018-07-20 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2020-11

CONDITIONS: Very Low Birth Weight Infant
Keywords: intravenous fat emulsions; preterm infants
MeSH Terms: interventions — Fat Emulsions, Intravenous; soybean oil, phospholipid emulsion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Begins treatment with 0.5 g/kg per day of 20% Intravenous Lipid Emulsion (IVLE) after birth if the birth weight is less or equal 1000g or 1 g/kg per day if birth weight is more than 1000g. The IVLE dose in this group will be increased by 0.5 g/kg per day daily until reaching 3 g/kg per day.
- experimental group (Experimental): The experimental group will begin treatment with 2 g/kg per day of 20% Intravenous Lipid Emulsion after birth.
  The dose of IVLE will be increased directly from 2 to 3 g/kg per day the next day in this group.
  Interventions: Other: Intravenous lipid emulsion

INTERVENTIONS:
Other: Intravenous lipid emulsion — using higher dose of IV lipids after birth
  Other Names: Intralipid
  Arms: experimental group

SUMMARY:
Provision of high and early fat intake may help to reduce the amount of postnatal weight loss in Very Low Birth Weight Infants. It may also help utilize the high amount of protein that is currently recommended to these premature babies. Also, we expect babies who get this appropriate intake to regain their birth weight earlier than others who are on slow fat increase regimen.

DETAILED DESCRIPTION:
The recommendation of the Pediatric Societies of North America and Europe is that postnatal growth of preterm infants matches the in-utero growth rates of fetuses that remain in utero until full-term. Despite this long-standing recommendation, approximately 43% to 97% of very low birth weight (VLBW, less than 1500 g) infants grow slower than the estimated fetal growth velocity. This slow postnatal growth usually results in extra-uterine growth restriction (EUGR), defined as having a measured growth parameter (weight, length, or head circumference) that is less than 10th percentile of intrauterine growth expectation based on estimated postmenstrual age (PMA) in premature neonates at the time of hospital discharge.4 EUGR is associated with major morbidities such as bronchopulmonary dysplasia (BPD), retinopathy of prematurity (ROP) and impaired neurodevelopment.

Although the etiology of EUGR is multifactorial, inadequate nutrition plays a pivotal role. There are three critical stages of nutrition support in VLBW infants: (1) acute stage during the first 1-3 weeks after birth when infants are on parenteral nutrition, (2) intermediate period when infants are slowly advanced to full enteral nutrition (growing care stage), and (3) the post-discharge stage. Failure to provide adequate nutrition in the acute stage result in cumulative energy and protein deficits that is difficult to reverse in the second stage. Inadequate early postnatal nutrition results in excessive weight loss that cannot be explained by the physiologic contraction of body water alone. The regain of birth weight may need two to three weeks or even longer in preterm infants with excessive postnatal weight loss.

Newborn infants born at term normally lose 5-10% of their body weight in the first week of life due to contraction of extracellular water compartment. The proportion of weight loss is significantly higher in VLBW infants. Increased insensible water loss is widely considered as the main cause for additional weight loss in this population. Nevertheless, studies identified low energy intake to be a key driver to excessive weight loss. In fact, an earlier study showed that significant postnatal weight loss occurs mainly in infants whose energy intake is inadequate. A more recent epidemiologic study demonstrated similar postnatal growth trajectories with a minimal crossing of percentiles after the initial weight loss regardless of gestational age at birth. The growth trajectories for infants in that study had similar slopes and growth rates which indicate that proportion of postnatal weight loss is a lead cause for EUGR at discharge. Therefore, we speculate that decreasing the maximum percentage of initial weight loss in the acute stage would keep the preterm infant on a higher growth trajectory that is enough to reduce the incidence of EUGR.

Current fat provision regimen for preterm infants include starting parenteral lipid at 12-24 hours of age with 0.5-1 g/kg per day and advancing by 0.5 g/kg/day until reaching 3 g/kg per day. Using early (within one hour of birth) and higher (start at 2 g/kg per day and advance to 3g/kg per day once total fluid intake is increased to 80 ml/kg/day) parenteral fat intake could reduce the cumulative caloric deficit in the acute stage. Because of high-density energy in fat, higher parenteral fat intake will reduce the early energy deficit and enhance protein accretion. The first 2-3 weeks of life offer a critical window to limit postnatal nutritional and energy deficits. Recent study showed that higher energy and fat intakes during the first 2 weeks after birth are associated with a lower incidence of brain lesions and dysmaturation at term equivalent age in preterm neonates.

To date, studies of "early aggressive nutrition" in preterm infants have mainly focused on high protein intake to prevent protein catabolism. Nevertheless, provision of high protein intake without enough energy is unlikely to significantly reduce the early loss of protein and fat mass that had been accreted before birth.

ELIGIBILITY:
Inclusion Criteria:

1. Preterm infants born with birth weight < 1500 g
2. Appropriate for gestational age (AGA)
3. Anticipated duration of PN for >7 days

Exclusion Criteria:

1. Infants with congenital anomalies
2. Infants with suspected inborn errors of metabolism or family history of inborn error of metabolism
3. Infants with suspected or confirmed biliary atresia
4. Infants born small for gestational age (SGA)
5. Confirmed early sepsis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2019-07-08 (Actual); Study Completion 2019-10-19 (Actual)

PRIMARY OUTCOMES:
The maximum percentage of weight loss | Until patient regains birth weight, on average within 14 days
  (birth weight-lowest postnatal weight)/birth weight× 100).

CONTACTS AND LOCATIONS:
Overall Officials: Belal Alshaikh, MD,MSc, Principal Investigator — University of Calgary
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alburaki W, Yusuf K, Dobry J, Sheinfeld R, Alshaikh B. High Early Parenteral Lipid in Very Preterm Infants: A Randomized-Controlled Trial. J Pediatr. 2021 Jan;228:16-23.e1. doi: 10.1016/j.jpeds.2020.08.024. Epub 2020 Aug 13. PMID 32798567

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-12-27): https://cdn.clinicaltrials.gov/large-docs/74/NCT03594474/Prot_SAP_000.pdf
  • Informed Consent Form (2017-12-27): https://cdn.clinicaltrials.gov/large-docs/74/NCT03594474/ICF_001.pdf